CLINICAL TRIAL: NCT04797572
Title: CALIBRATE TRIAL: a Prospective, Single Arm Investigational Clinical Trial Evaluating Safety and Performance of the Free Margin Cusp Sizer During Aortic Valve Repair Surgery
Brief Title: Clinical Evaluation of the Free Margin Cusp Sizer (CALIBRATE)
Acronym: CALIBRATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALIBRATE TRIAL01; 2020-14DEC/619 (Other: Ethics Committee, Cliniques Universitaires Saint-Luc, UCL)
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Aortic Valve Regurgitation; Aortic Root Aneurysm
Keywords: aortic valve repair; Valve sparing surgery; Trileaflet aortic valve
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Root Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treated group (Other): Patients in whom the free margin cusp sizer will be used to measure the free margin of the three leaflets of the aortic valve during aortic valve repair.
  Interventions: Device: Free Margin Cusp Sizer

INTERVENTIONS:
Device: Free Margin Cusp Sizer — The free margin cusp sizer will be used during aortic valve repair and sparing procedures as a caliper to measure the aortic valve free margin length.

SUMMARY:
The objective of this study is to investigate safety and performance of the Free Margin Cusp sizer. The device will be used during aortic valve repair and sparing procedures as a caliper to measure the aortic valve free margin length at different stages of the procedure. The patient will be followed for one year clinically (at 1, 2, 6 and 12 months) and by echocardiography (at 6 and 12 months) to assess aortic valve function.

DETAILED DESCRIPTION:
Goal of the study :

The objective of this study is to study the safety and reliability of a new surgical instrument, the "Free Margin Cusp Sizer" (patented device). The measuring instrument will be used during aortic valve repair procedures to measure the length of the free edge of the aortic cusps.

State of the art :

Currently, aortic valve repair is done by visual estimation and requires a great level of experience from the surgeon. We proposed to develop an objective cusp repair technique based on the measurement of the free edge by a dedicated sizer. The measuring instrument will give the objective difference in millimeters between the normal cusp and the one with prolapse. This will then be quantitatively plicatured to correct its excess length. This new technique will allow less experienced surgeons or those in the process of learning objective guidance of valve repair. The objective measure of the free edge length may also orient the sizing of the Dacron graft used for valve sparing root replacement.

Study evaluation criteria:

* Hospital mortality (mortality at 30 days), MACCE at one year: mortality, cerebrovascular accident or transient ischemic attack, major hemorrhage, cardiac reoperation
* Echocardiographic results at discharge from hospital and at 6 months or one year

Material and methods:

* Single-center, prospective, non-randomized study
* Patient source: Patients operated for aortic valve repair or aortic valve sparing surgery at Cliniques Universitaires Saint-Luc (CUSL), Brussels
* Number of patients to be included: 120, study duration: 6,5 years, inclusion period: 5,5 years, follow-up:

  1 year
* Inclusion criteria: patient with a tricuspid aortic valve operated electively for aortic valve insufficiency or dilation of the ascending aorta
* Exclusion criteria: acute aortic dissection, diffuse aortic valve calcification, endocarditis, bicuspide, unicuspid or quadricuspid aortic valve, patient under 18 and over 80

Data acquisition and patient follow-up:

The examinations carried out within the framework of this study are the same as those carried out routinely during the preoperative cardiac assessment and clinical follow-up after aortic valve repair:

* Preoperative cardiovascular examination including TTE (transthoracic ultrasound) / TEE (transesophageal ultrasound)
* Intraoperative TEE pre and post aortic valve repair
* TTE at discharge
* TTE between 6 months and one year postoperatively
* 1 month post-operative consultation (outpatient surgery)
* Consultation 1 to 2 months postoperative (referring cardiologist)
* Consultation 6-12 months postoperative (referring cardiologist) (if necessary, phone contact with the patient at 12-14 months)

ELIGIBILITY:
Inclusion Criteria:

* Patients with Tricuspid Aortic Valve (TAV) operated electively for aortic valve regurgitation and or ascending aorta dilatation.

Exclusion Criteria:

* Acute aortic dissection;
* Diffuse aortic valve calcification;
* AV endocarditis;
* Bicuspid, unicuspid or quadricuspid aortic valves;
* Patients under the age of 18 years;
* Patients above the age of 80 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative aortic valve (AV) damage | 30 days
  Aortic valve damage caused by the cusp sizer (cusp tear or perforation), rate of conversion from AV repair to AV replacement due to the use of the cusp sizer
Hospital mortality | 30 days
  Patient Survival status at 30 days after surgery
Major adverse cardiac and cerebrovascular events (MACCE) | one year
  Mortality, stroke or transient ischemic attack, major bleeding, cardiac reintervention
Aortic valve function | One year
  Aortic valve regurgitation and transvalvular gradient by transthoracic echocardiography

SECONDARY OUTCOMES:
Pre-repair free margin length | Intraoperative
  Length of the 3 leaflets free margin before aortic valve repair

CONTACTS AND LOCATIONS:
Overall Officials: Laurent de kerchove, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Kerchove L, Momeni M, Aphram G, Watremez C, Bollen X, Jashari R, Boodhwani M, Astarci P, Noirhomme P, El Khoury G. Free margin length and coaptation surface area in normal tricuspid aortic valve: an anatomical study. Eur J Cardiothorac Surg. 2018 May 1;53(5):1040-1048. doi: 10.1093/ejcts/ezx456. PMID 29253123
- [Background] Tamer S, Mastrobuoni S, van Dyck M, Navarra E, Bollen X, Poncelet A, Noirhomme P, Astarci P, El Khoury G, de Kerchove L. Free margin length and geometric height in aortic root dilatation and leaflet prolapse: implications for aortic valve repair surgery. Eur J Cardiothorac Surg. 2020 Jan 1;57(1):124-132. doi: 10.1093/ejcts/ezz132. PMID 31089691